CLINICAL TRIAL: NCT00822029
Title: Use of Oral Bisphosphonates in the Treatment of Osteoporosis of Non-walking Children With Cerebral Palsy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: only 2 patients inclued and Study Principal Investigator has left the hospital
Sponsor: Department of Clinical Research and Innovation (Other)
Responsible Party: Sponsor-Investigator, Department of Clinical Research and Innovation, Departement of clinical research and innovation (drc), Centre Hospitalier Universitaire de Nice
Organization: Centre Hospitalier Universitaire de Nice (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006-005678-36
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2011-11

CONDITIONS: Osteoporosis; Cerebral Palsy
MeSH Terms: conditions — Osteoporosis; Cerebral Palsy | interventions — Alendronate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): FOSAMAX (oral bisphosphonate)
  Interventions: Drug: FOSAMAX
- 2 (Placebo Comparator): PLACEBO
  Interventions: Other: PLACEBO

INTERVENTIONS:
Drug: FOSAMAX — patient receiving one tablet (oral use) 70 mg Fosamax by week
  Arms: 1
Other: PLACEBO — patient receiving one tablet (oral use) placebo by week
  Arms: 2

SUMMARY:
It is a double blind randomized study aiming at estimating the efficiency of oral bisphosphonates on the decrease of osteoporosis by comparing the evolution of densitometric values between two groups of children (treatment versus placebo).

DETAILED DESCRIPTION:
In non walking children with cerebral palsy, osteoporosis is responsible for bone pains and iterative fractures. Classical treatments include physiotherapy, assisted verticalisation by orthesis and correct feeding with vitamin D and calcium supplementation. Yet this isn't always sufficient and isn't always possible.

Bisphosphonates, which have been used for years in the treatment of post-menopausic osteoporosis or of osteogenesis imperfecta in children, can turn out to be very useful for non-walking children with cerebral palsy.

Studies have been published since 1994 in this indication with encouraging results. Cyclic intravenous administration of bisphosphonates every 3 months showed an objective increase in bone density and a decrease in pains and fractures after one year of treatment. Cyclic intravenous administration nevertheless requires the use of an implanted chamber and iterative hospitalizations. Oral administration should allow to treat these children, who already have many treatments, in a simpler way.

The study will concern 40 non-walking children with cerebral palsy aged over 10 years.

ELIGIBILITY:
Inclusion Criteria:

* non-walking children with cerebral palsy
* weight > to or = 20 kg
* aged between 10 to 18 years old
* with a Z-score (spinal and / or femoral) <-2 DS
* with a good dental status
* capable of holding the seated or half seated position for 30 minutes
* capable of filling the study questionary
* with negative blood pregnancy tests on inclusion for pubescent girls
* Using valid contraception means (condoms, oral contraception) for pubescent girls for the whole study duration and 6 months after the end of the study
* affiliated to the social security regimen

Exclusion Criteria:

* history of spine arthrodesis with osteosynthesis
* gastro-oesophageal reflux
* oesophagal disease or any factor leading to a delaying or slowing the oesophagal transit (such as stenosis or achalasy)
* severe difficulties in swallowing
* renal failure
* history of uveitis
* hypersensibility to alendronate or to one of its excipients (microcristalline cellulose, lactose anhydre, croscarmellose sodium, magnesium stearate)
* deficiency in calcium or in vitamine D
* calcium malabsorption
* hereditary galactose intolerance, congenital galactosemia, glucose and galactose malabsorption syndrome
* evolutive affection of the upper gastro-intestinal tract such as dysphagia (other than neurological), gastritis, duodenitis, gastro-duodenal ulcers (or with history of ulcers in the previous year), evolutive gastro-intestinal bleeding or history of surgery of the upper gastro-intestinal tract (gastrostomy in particular)
* history of necrosis of the maxillar bone or of uncovering of the bone or of cicatrisation delay after a dental surgery
* emancipated minor
* prior treatment with bisphosphonates
* inclusion in another clinical research study

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2009-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
To estimate the efficiency of oral bisphosphonates on the decrease of osteoporosis assessed by osteodensitometry. | one year

SECONDARY OUTCOMES:
To estimate the improvement of the biological and clinical consequences (bone pains and fractures) of osteoporosis. To estimate the improvement of the quality of life To estimate the tolerance of oral bisphosphonates. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Jacques GRIFFET, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- Chirurgie Infantile - Hôpital ARCHET, Nice, France